CLINICAL TRIAL: NCT02578797
Title: An Open-Label Phase 1b QT/QTc Study of JNJ-56021927 (ARN-509) in Subjects With Castration-Resistant Prostate Cancer
Brief Title: A JNJ-56021927 (ARN-509; Apalutamide) QT/QTc Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108049; 2015-004044-19 (EudraCT Number); 56021927PCR1019 (Other: Aragon Pharmaceuticals, Inc)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Castration-Resistant Prostate Cancer
Keywords: Castration-Resistant Prostate Cancer (CRPC); Prostatic Neoplasms; Genital Diseases, Male; Genital Neoplasms, Male; Neoplasms; Neoplasms by Site; Prostatic Diseases; Urogenital Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Genital Diseases, Male; Genital Neoplasms, Male; Neoplasms; Neoplasms by Site; Prostatic Diseases; Urogenital Neoplasms | interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Apalutamide (Experimental): Prostate Cancer participants will receive the study drug on an outpatient basis except for Cycle 1 (Day 1 and Day 2) and Cycle 3 (Day 1), when intake must occur at study site under overnight fasted conditions.
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Apalutamide — Study drug will be administered orally at a dose level of 240 mg daily (4 x 60 mg tablets) in treatment cycles of 28 days.

SUMMARY:
The purpose of this study is to determine whether daily treatment with apalutamide affects the ventricular repolarization in participants with Castration-Resistant Prostate Cancer (CRPC)

DETAILED DESCRIPTION:
This is an open-label (a study in which the drug, procedure is known to participant and investigator), multicenter, Phase 1b study to investigate the effect of apalutamide on ventricular repolarization at a dose level of 240 milligram (mg daily). Approximately 42 participants with high-risk non-metastatic prostate cancer (NM-CRPC), defined as having a prostate specific antigen (PSA) doubling time less than or equal to (<=) 10 months, or participants with metastatic CRPC will be enrolled. The study consists of a 28-day Screening Phase, a Treatment Phase and a Follow-up Phase. In the Treatment Phase the study drug will be administrated in cycles of 28 days and the participants will be monitored for safety (including cardiac safety) and pharmacokinetics of the study drug. Adverse Events will be monitored throughout the study and in the Follow-up Phase until 30 days after the last dose of study drug. All participants will continue on study until disease progression, withdrawal of consent, lost to follow-up, the occurrence of unacceptable toxicity, the participant is no longer receiving clinical benefit in the opinion of the investigator, or termination of the study by the sponsor. Upon discontinuation of study drug, the participants will return for an End-of-Treatment (EoT) visit no later than 30 days after their last dose. The end of the study corresponds to the clinical cutoff and end of data collection.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adenocarcinoma of the prostate; either non-metastatic castrate resistant prostate cancer (NM-CRPC) with high risk disease (defined as PSA Doubling time equal or less than (<=) 10 months) or metastatic CRPC
* Be surgically or medically castrated with testosterone levels of less than (<) 50 nanogram per deciliter
* If treated with a gonadotropin releasing hormone analog (ie, patient who has not undergone bilateral orchiectomy), then this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study
* Electrocardiogram (ECG) showing a QT interval corrected for heart rate, using Fridericia formula (QTcF) <= 470 milliseconds (based on the average of a triplicate ECG set collected during the screening visit)
* Left ventricular ejection fraction (LVEF) of more than 45% as determined by multiple uptake gated acquisition (MUGA) or echocardiography at the screening visit

Exclusion Criteria:

* Abnormal cardiac function at screening
* Known brain metastases
* Has received an investigational drug within 4 weeks, or within a period < 10 times the drug's half-life, whichever is longer, of Cycle 1 Day 1
* Has received chemotherapy or immunotherapy for the treatment of prostate cancer within 4 weeks of Cycle 1 Day 1
* Prior treatment with enzalutamide and apalutamide
* Use of therapies that must be discontinued or substituted within at least 4 weeks prior to Cycle 1 Day 1 including medications to lower seizure threshold, inducing/inhibiting metabolizing enzymes or prolonging the QT interval
* History or condition that may predispose to seizures, or evidence of severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events within 12 months prior to Cycle 1 Day 1, New York Heart Association (NYHA) Class II to IV heart disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
QTc Fridericia (QTcF) parameter | Day-1 and Day 1 (Cycle 1) and Day 1 (Cycle 3)
  Mean change from baseline in QTcF as measured based on triplicate electrocardiograms extracted from continuous 12-lead Holter monitor recordings after study drug intake.

SECONDARY OUTCOMES:
Electrocardiographic parameters (HR, RR, PR, and QRS) | Day-1 and Day 1 (Cycle 1) and Day 1 (Cycle 3)
  A change from time-matched baseline measurements in HR, PR, RR and QRS interval will be determined on Day -1, Day 1 and Day 3
Electrocardiographic parameters (QT) | Day-1 and Day 1 (Cycle 1) and Day 1 (Cycle 3)
  QT interval on a surface ECG will be corrected for heart rate using Bazett formula (QTcB) and study-specific Power (QTcP) if appropriate at each treatment period.
Electrocardiographic parameters T- and U-wave morphology | Day-1 and Day 1 (Cycle 1) and Day 1 (Cycle 3)
  Number and percentage of participants with changes from baseline
Plasma concentrations apalutamide (and its active metabolite JNJ-56142060) | Day-1, Day 1 and Day 2 (Cycle 1) and Day 1 (Cycle 3)
  Blood samples will be taken following dose administration.
Number of participants with Adverse Events | Day-1, Day 1 and Day 15 (Cycle 1); Day 1 and Day 15 (Cycle 2) and Day 1 (Cycle 3).
  Participants will be monitored for safety during the Screening and Treatment Phases, and up to 30 days after the last dose of study drug. From Cycle 4 onward collection of Adverse Events (AEs) will be limited to Grade 3 or higher and all Serious AEs from the remainder of the study.
Pharmacokinetic parameter area under the plasma drug concentration-time curve (AUC) from time 0 to 24 hours | Day 1 and Day 2 (Cycle 1) and Day 1 (Cycle 3)
  The AUC(0-24h) is the area under the plasma concentration-time curve from time 0 to time 24 hours after dosing.
Pharmacokinetic parameter maximum concentration observed (Cmax) | Day 1 and Day 2 (Cycle 1) and Day 1 (Cycle 3)
  The Cmax is the maximum observed plasma concentration.
Pharmacokinetic parameter time to reach Cmax (tmax) | Day 1 and Day 2 (Cycle 1) and Day 1 (Cycle 3)
  The tmax is the time to reach the maximum observed plasma concentration.
Pharmacokinetic parameter minimum observed plasma concentration (Cmin) | Cmin will only be collected on Day 1, Cycle 3
  The Cmin is the minimum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Greenville, South Carolina, United States
- Montreal, Quebec, Canada
- Chisinau, Moldova
- Rotterdam, Netherlands
- Sutton, United Kingdom